CLINICAL TRIAL: NCT05329662
Title: Evaluation of Autologous Adipose Tissue-derived Mesenchymal Stem Cell Efficacy for the Treatment of Sexual Function Impairment in Female
Brief Title: Adipose Tissue-derived Mesenchymal Stem Cell (AD-MSC) Therapy for the Treatment of Sexual Function Impairment in Female
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vinmec Research Institute of Stem Cell and Gene Technology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: ISC.21.73
Record Dates: First submitted 2022-04-07; First posted 2022-04-15 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Sexual Dysfunction Female
Keywords: sexual dysfunction Female; adipose mesenchymal stem cell; reproductive hormones

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AD-MSCs infusions, then Placebo (Active Comparator): Patients in group A will receive two autologous AD-MSC administrations on day 0 and day 90 ± 7
  Interventions: Biological: Autologous adipose-derived mesenchymal stem cell administration for female with sexual functional deficiency
- Placebo, then AD-MSCs infusions (Placebo Comparator): Patients in group B will receive two autologous AD-MSC administrations on day 180 ± 14 and day 270 ± 14
  Interventions: Biological: Autologous adipose-derived mesenchymal stem cell administration for female with sexual functional deficiency

INTERVENTIONS:
Biological: Autologous adipose-derived mesenchymal stem cell administration for female with sexual functional deficiency — * Patients in the two groups will receive two autologous AD-MSC administrations: the group A on day 0 and day 90 ± 7; the group B on day 180 ± 14 and day 270 ± 14.
  * Dose: 1.0 x 106 cells/kg patient bodyweight.
  * Route: intravenous infusion
  ADSCs were collected after the third passage. On the day of transplantation, the ADSCs were harvested, washed twice with NaCl 0.9%, counted and resuspended in NaCl 0.9% in a total volume of 20 ml. Each participant received a dose of 1x10^6 cells/kg body weight infused through the intravenous route within 30 minutes before being discharged after 24 hours

SUMMARY:
Hormones are a chemical substance synthesized and secreted by endocrine gland. Several vital hormones, including Mullerian hormone (AMH), follicle-stimulating hormone (FSH), and Estradiol (E2), play crucial roles in regulating female sexual function.- Hormone therapy is used to treat female hormone deficiency and results in a significant improvement, but long-term use increases cardiovascular disease or cancer risk. Other treatments do not give apparent results. Therefore, it is necessary to develop new and effective treatments to achieve the requirements of improving health in general and sexual health in particularly in women. AD-MSCs have been widely used as autologous and allogeneic stem cell sources to treat numerous disease recently, and they have been proven to be safe. The phase I trial showed that administration of autologous AD-MSCs at the dose of 1.0 x 10^6 cells/kg patient bodyweight was safe for patients with sex hormone deficiency. The therapy introduced potential improvement in sexual and general quality of life indicating by the increased FSFI. Therefore, this phase II trial to evaluate efficiency of autologous adipose tissue-derived mesenchymal stem cells therapy in treatment of female patients with sexual function impairment.

DETAILED DESCRIPTION:
Hormones are a chemical substance synthesized and secreted by endocrine gland. They are used by multicellular organism to organize, coordinate, and regulate multiple functions of cells and tissues in the body. They are considered as chemical messenger molecules that send signals from one cell to another within or between various body parts. Hormones are responsible for regulating many physiological processes and behavioral activities such as growth and development of the body, metabolism, homeostasis of intracellular and extracellular fluid, and reproduction. Several vital hormones, including Mullerian hormone (AMH), follicle-stimulating hormone (FSH), and Estradiol (E2), play crucial roles in regulating female sexual function. The phase I clinical study named " Single-group, open-label clinical trial, evaluating the safety and efficacy of adipose tissue-derived mesenchymal stem cell therapy for early sex hormone deficiency in middle-aged people" showed that AD-MSC therapy for patients with hormone deficiency is safe, can improve the sexual quality of life in both men and women. A significant statistical increase of testosterone levels was observed in male patients at 3-month, 6-month and 12-month. In female patients, the FSFI was 20.70 at baseline and increased to 27.1 at 12 months after AD-MSC infusion (p<0.05). There were no significant changes in AMH, FSH, or E2 infusion compared to baseline in the 16 enrolled patients. Within those under 45 years old, FSH and E2 tended to increase at 3 months after ADSC infusion and decreased at the follow-up after 6 and 12 months. Therefore, this phase II trial to evaluate efficiency of autologous adipose tissue-derived mesenchymal stem cells therapy in treatment of female patients with sexual function impairment.

ELIGIBILITY:
Inclusion Criteria:

* Women who are 40 - 50 years of age or older and have not gone through menopause according to Stages of Reproductive Aging Workshop (STRAW) 2011
* The last menstrual period before participating in the study at least 2 months or more
* FSH, Estrogen above the menopause:
* + FSH > 40 mIU/mL
* + Estradiol < 30 pg/mL
* (tested between the 2nd and the 4th day of the menstrual cycle)
* FSFI < 26.55 ± signs of decline in sexual or reproductive functions such as symptoms of premenopausal such as hot flashes, excessive sweating, headaches
* Normal liver function
* Normal kidney function
* Normal cardiovascular function
* No active bacterial, fungal and viral (HIV, HBV, HCV, syphilis) infections
* Provide written informed consent

Exclusion Criteria:

* Previous surgery to remove gonads
* No sexual activity
* Diagnosed with cancer and is being or has not been treated
* Had an organ transplant
* Has congenital malformations related to the gonads
* Chronic disease such as: Diabetes, hypopituitarism, adrenal insufficiency, blood pressure unresponsive to treatment, etc
* Any active autoimmune diseases
* Being diagnosed with heart failure, kidney failure, liver failure, respiratory failure, history of cerebral infarction, myocardial infarction, Alzheimer's
* Hypothyroidism or hyperthyroidism
* Any active autoimmune diseases
* Any clinically significant blood coagulation disorders.
* History of allergic reaction to anesthetic agents and antibiotics
* Using hormone therapy within the last 2 weeks or want to use these drugs during the study period
* Planning to become pregnant during the study period
* using hormonal contraceptives
* Absence of menstruation for at least 12 months
* Mental illness, inability to communicate, inability to answer the interview questions correctly

Ages: 40 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 130 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change of Follicle-stimulating hormone (FSH) hormone level | 1 month, 3 months, 6 months, 12 months after the first UCMSC infusion
  FSH stimulates granulosa cells in the ovarian follicles to synthesize aromatase, which converts androgens produced by the thecal cells to estradiol. FSH peaks at the same time as the LH surge that causes ovulation. FSH then remains low throughout the luteal phase, preventing the development of new follicles. FSH levels is measured in the serum sample.
Change of Estradiol (E2) hormone level | 1 month, 3 months, 6 months, 12 months after the first UCMSC infusion
  Estrogen is a steroid hormone associated with the female reproductive organs and is responsible for the development of female sexual characteristics.
Change in Quality of life using Female Sexual Function Index - FSFI questionaires | 1 month, 3 months, 6 months, 12 months after the first UCMSC infusion
  The FSFI questionnaire consists of 19 close-ended questions related to sexual activity within the 4 weeks prior to the examination. Points are assigned for each answer (1-5 and 0-5 for questions 1-2 and questions 3-19, respectively), the sum of the scores for the domain is multiplied by the domain factor, the six domain scores are added up, and the total score may vary from 2.0 to 36.0 points.
Change in Quality of life using The Utian Quality of life Scale | 1 month, 3 months, 6 months, 12 months after the first UCMSC infusion
  The UQOL is the first pure QOL measure of this new generation of instruments that can be applied to a menopausal population. Items are scaled using a Likert-type 1 to 5 rating.

SECONDARY OUTCOMES:
The safety of AD MSC therapy in the treatment of sexual function impairment in female | 1 month, 3 months, 6 months, 12 months after the first UCMSC infusion
  The frequency and severity of AEs and SAEs during the intervention and within 12 months after the first cell administration.

CONTACTS AND LOCATIONS:
Overall Officials: Tan Sinh Nguyen, PhD, Principal Investigator — Vinmec Times City International Hospital
Locations (1):
- Vinmec Research Institute of Stem Cell and Gene Technology, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No